CLINICAL TRIAL: NCT04945317
Title: Rapid Onsite Cytopathologic Evaluation for Improved Molecular Marker Testing Via Endobronchial Ultrasound Bronchoscopy - A Randomized Controlled Trial
Brief Title: ROSE for Improved Molecular Marker Testing Via EBUS
Acronym: ROSE/NoROSE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00162151
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Endobronchial ultrasound (EBUS); Rapid on-site evaluation (ROSE)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Multi-center non-blinded randomized controlled trial (presence or absence of trained cytotechnologist providing on-site cytopathology feedback to bronchoscopist).
Masking Description: blinding not possible given nature of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ROSE clot arm (Other): Presence of trained cytotechnologist providing on-site cytopathology feedback to bronchoscopist. Sample prepared as tissue clot.
  Interventions: Other: ROSE (presence of cytotech) & tissue clot sample
- NO-ROSE clot arm (Other): Absence of trained cytotechnologist providing on-site cytopathology feedback to bronchoscopist. Sample prepared as tissue clot.
  Interventions: Other: NO-ROSE (absence of cytotech) & tissue clot sample
- ROSE liquid arm (Other): Presence of trained cytotechnologist providing on-site cytopathology feedback to bronchoscopist. Sample prepared as liquid.
  Interventions: Other: ROSE (presence of cytotech) & liquid prep
- NO-ROSE liquid arm (Other): Absence of trained cytotechnologist providing on-site cytopathology feedback to bronchoscopist. Sample prepared as
  Interventions: Other: NO-ROSE (absence of cytotech) & liquid prep

INTERVENTIONS:
Other: ROSE (presence of cytotech) & liquid prep — Standard of care EBUS will include presence of trained cytotechnologist providing on-site cytopathology feedback to bronchoscopist during the procedure. Sample is liquid.
  Arms: ROSE liquid arm
Other: NO-ROSE (absence of cytotech) & liquid prep — Standard of care EBUS will NOT include presence of trained cytotechnologist providing on-site cytopathology feedback to bronchoscopist during the procedure. Sample is liquid.
  Arms: NO-ROSE liquid arm
Other: ROSE (presence of cytotech) & tissue clot sample — Standard of care EBUS will include presence of trained cytotechnologist providing on-site cytopathology feedback to bronchoscopist during the procedure. Sample is a tissue clot.
  Arms: ROSE clot arm
Other: NO-ROSE (absence of cytotech) & tissue clot sample — Standard of care EBUS will NOT include presence of trained cytotechnologist providing on-site cytopathology feedback to bronchoscopist during the procedure. Sample is a tissue clot.
  Arms: NO-ROSE clot arm

SUMMARY:
This research study is being done to compare two ways to conduct bronchoscopic biopsy of lymph nodes and other structures in the chest (i.e. the presence or absence of an on-site cytotechnologist performing a limited microscopic evaluation to provide non-binding feedback on specimen adequacy in real time during the procedure).

DETAILED DESCRIPTION:
Endobronchial ultrasound (EBUS) is a highly safe and effective bronchoscopic procedure that can achieve diagnostic yields of over 90% for lung cancer - similar to those with the more-invasive surgical mediastinoscopy - with EBUS enjoying the advantage of a near 0% complication rate in several large studies. This has led to EBUS becoming the procedure of choice for mediastinal staging of lung cancer. Increasingly, bronchoscopists are being asked to perform EBUS not only for lung cancer staging but also for tissue acquisition for molecular markers to assess for mutations that can be treated with biologic therapy. However, a frequently encountered clinical scenario is that while an EBUS is diagnostic for lung cancer, it is non-diagnostic for molecular testing because of an insufficient amount of tissue material being collected. According to multiple studies, the "molecular yield" for EBUS in lung cancer can range from 74-82%. These studies have not specifically looked at adequacy of biomarkers, which could be distinctly different considering that evaluation of biomarkers requires more tissue for next generation sequencing (NGS). Currently, Johns Hopkins Hospital uses NGS as standard of care for identifying mutations associated with malignant cells. NGS analysis, which is usually reported as a percentage of cells that express one of many biomarkers currently being tested as standard of care, is performed via immunohistochemistry (IHC), necessitating the presence of a sufficiently cellular material with >100 tumor cells for reliable quantitative characterization. To the investigator's knowledge, the rates of NGS biomarker sufficiency have not been prospectively analyzed to date.

Rapid on-site evaluation (ROSE) is an optional step during EBUS bronchoscopy in which an on-site cytotechnologist performs a limited microscopic evaluation to provide non-binding feedback on specimen adequacy in real time during the procedure. The cytotechnologist can also aid specimen processing e.g. through creation of a "tissue clot" in addition to use of the more standard liquid-based medium. At Johns Hopkins, EBUS procedures are routinely performed both with and without ROSE since the presence or absence of ROSE during EBUS has not been shown to impact diagnostic yield or procedural safety. However, its impact on NGS biomarker sufficiency has not been tested to the investigator's knowledge.

This study aims to investigate whether ROSE can impact NGS biomarker sufficiency by assisting the bronchoscopist in obtaining adequate tissue from the appropriate site. The hypothesis is that ROSE will decrease the rate of insufficient tumor tissue to permit NGS biomarker testing.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients or outpatients >18 years old
* Capable of informed consent
* Known or suspected non-small cell lung cancer (NSCLC)
* Referred to the interventional pulmonary team at Johns Hopkins Hospital (JHH), Johns Hopkins Bayview Medical Center (JHBMC), or other participating sites for tissue sampling of a hilar/mediastinal lymph node or another lesion accessible by convex-probe (CP) EBUS

Exclusion Criteria:

* Refuse participation
* Standard contraindications to EBUS and bronchoscopy in general: bleeding disorders, antiplatelet or anticoagulant usage, high fraction of inspired oxygen (FiO2) requirement, and clinical instability
* Pregnant women
* Cytotechnologist not available at the time of screening, enrollment, or randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of NGS biomarker testing attempts | within 60 days of procedure
  NGS biomarker sufficiency - percentage of NGS biomarker testing attempts that were successful due to sufficient tissue

SECONDARY OUTCOMES:
Level of Programmed Cell Death Protein 1 (PD-1) | within 60 days of procedure
  PD-1 sufficiency - amount of the protein "Programmed Cell Death Protein 1" (PD-1) expressed on immune cells = 500 cells/20% cellularity
Number of targets | During Procedure
  Number of targets (including lymph node stations, other lesions) sampled per EBUS
Number of passes (ROSE arms only) | During Procedure
  Number of passes taken from the target site
Number of secondary procedures | During Procedure
  Number of secondary procedures performed (such as radial EBUS, navigational bronchoscopy)
Need for repeat EBUS or another procedure | Within 30 days of procedure
  Need for repeat EBUS or another procedure due to non-diagnostic or insufficient sample during a 30-day follow up period (binary value: yes/no)
Procedure time | During Procedure
  Procedure time (measured in minutes)
Number of Procedural complications | Within 7 days of the procedure
  Procedural complications observed during a one-week follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, DO, MBA, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Northwestern Medicine, Chicago, Illinois
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Medical University of South Carolina (MUSC), Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annema JT, van Meerbeeck JP, Rintoul RC, Dooms C, Deschepper E, Dekkers OM, De Leyn P, Braun J, Carroll NR, Praet M, de Ryck F, Vansteenkiste J, Vermassen F, Versteegh MI, Veselic M, Nicholson AG, Rabe KF, Tournoy KG. Mediastinoscopy vs endosonography for mediastinal nodal staging of lung cancer: a randomized trial. JAMA. 2010 Nov 24;304(20):2245-52. doi: 10.1001/jama.2010.1705. PMID 21098770
- [Background] Varela-Lema L, Fernandez-Villar A, Ruano-Ravina A. Effectiveness and safety of endobronchial ultrasound-transbronchial needle aspiration: a systematic review. Eur Respir J. 2009 May;33(5):1156-64. doi: 10.1183/09031936.00097908. PMID 19407050
- [Background] Anantham D, Koh MS, Ernst A. Endobronchial ultrasound. Respir Med. 2009 Oct;103(10):1406-14. doi: 10.1016/j.rmed.2009.04.010. Epub 2009 May 15. PMID 19447014
- [Background] Silvestri GA, Gonzalez AV, Jantz MA, Margolis ML, Gould MK, Tanoue LT, Harris LJ, Detterbeck FC. Methods for staging non-small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e211S-e250S. doi: 10.1378/chest.12-2355. PMID 23649440
- [Background] Sakakibara R, Inamura K, Tambo Y, Ninomiya H, Kitazono S, Yanagitani N, Horiike A, Ohyanagi F, Matsuura Y, Nakao M, Mun M, Okumura S, Inase N, Nishio M, Motoi N, Ishikawa Y. EBUS-TBNA as a Promising Method for the Evaluation of Tumor PD-L1 Expression in Lung Cancer. Clin Lung Cancer. 2017 Sep;18(5):527-534.e1. doi: 10.1016/j.cllc.2016.12.002. Epub 2016 Dec 22. PMID 28111119
- [Background] Oezkan F, Khan A, Zarogoulidis P, Hohenforst-Schmidt W, Theegarten D, Yasufuku K, Nakajima T, Freitag L, Darwiche K. Efficient utilization of EBUS-TBNA samples for both diagnosis and molecular analyses. Onco Targets Ther. 2014 Nov 10;7:2061-5. doi: 10.2147/OTT.S72974. eCollection 2014. PMID 25419143
- [Background] Jurado J, Saqi A, Maxfield R, Newmark A, Lavelle M, Bacchetta M, Gorenstein L, Dovidio F, Ginsburg ME, Sonett J, Bulman W. The efficacy of EBUS-guided transbronchial needle aspiration for molecular testing in lung adenocarcinoma. Ann Thorac Surg. 2013 Oct;96(4):1196-1202. doi: 10.1016/j.athoracsur.2013.05.066. Epub 2013 Aug 21. PMID 23972930
- [Background] Yung RC, Otell S, Illei P, Clark DP, Feller-Kopman D, Yarmus L, Askin F, Gabrielson E, Li QK. Improvement of cellularity on cell block preparations using the so-called tissue coagulum clot method during endobronchial ultrasound-guided transbronchial fine-needle aspiration. Cancer Cytopathol. 2012 Jun 25;120(3):185-95. doi: 10.1002/cncy.20199. Epub 2011 Dec 5. PMID 22144401
- [Background] Oki M, Saka H, Kitagawa C, Kogure Y, Murata N, Adachi T, Ando M. Rapid on-site cytologic evaluation during endobronchial ultrasound-guided transbronchial needle aspiration for diagnosing lung cancer: a randomized study. Respiration. 2013;85(6):486-92. doi: 10.1159/000346987. Epub 2013 Apr 3. PMID 23571718